CLINICAL TRIAL: NCT06871787
Title: Evaluation of Bowel Anastomoses During Gynecologic Oncology Surgery Using Near-Infrared Fluorescence Imaging With Indocyanine Green
Brief Title: Near-Infrared Fluorescence Imaging With Indocyanine Green to Evaluate Bowel Anastomoses in Gynecologic Oncology Surgery
Acronym: INOCA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Atahan Toyran, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07.01.2025-3097444
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic Cancers; Ovarian Cancer; Endometrial Cancers; Cervical Cancers; Vulvar Cancer; Anastomotic Leaks
Keywords: Indocyanine Green; Near-Infrared Imaging; Bowel Anastomosis; Gynecologic Oncology; Anastomotic Complications; Perfusion Assessment
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Anastomotic Leak | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ICG Fluorescence Imaging Group (Experimental): Women undergoing gynecologic oncology surgery with bowel resection and anastomosis. Anastomotic perfusion will be evaluated intraoperatively using indocyanine green (ICG) enhanced near-infrared fluorescence imaging.
  Interventions: Drug: Indocyanine Green; Device: Near-Infrared Fluorescence Imaging System

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine green (ICG), administered intravenously at a dose of 2.5 mg/ml, will be used during surgery to evaluate bowel anastomosis perfusion through near-infrared fluorescence imaging.
Device: Near-Infrared Fluorescence Imaging System — A near-infrared fluorescence imaging device will be used intraoperatively to visualize indocyanine green (ICG) fluorescence, assessing the perfusion of bowel anastomoses during gynecologic oncology surgery.

SUMMARY:
The goal of this study is to evaluate if indocyanine green (ICG) fluorescence imaging helps reduce complications in bowel surgery performed during gynecologic cancer operations.

The main question it aims to answer is: Does using ICG fluorescence imaging during bowel anastomosis reduce the rate of complications such as leaks, infections, and abscesses within 30 days after surgery? Participants are women aged 18 and older undergoing surgery for gynecologic cancers (such as ovarian, uterine, cervical, or vulvar cancer). During surgery, investigators will inject ICG intravenously, then use a special near-infrared camera to see how well blood flows at the anastomosis site. The investigators will then decide if the reconnection is good enough or needs adjustment.

Researchers will record any complications within the first 30 days after surgery to understand if this imaging method helps reduce surgical risks.

DETAILED DESCRIPTION:
In gynecologic cancer surgeries, complete removal of the tumor often requires bowel resection (removal of part of the intestine). After resection, surgeons perform bowel anastomosis to restore gastrointestinal continuity. However, anastomosis can sometimes fail, leading to complications such as leaks, pelvic abscesses, or infections. Such complications significantly affect patient health, recovery, and outcomes.

Indocyanine green (ICG) is a dye approved by health authorities for clinical use. When injected into the bloodstream, it glows brightly under near-infrared (NIR) light, allowing investigators to visually assess blood flow in tissues during surgery. Good blood flow is critical for proper healing of the bowel reconnection.

This study aims to evaluate the effectiveness of using ICG-enhanced NIR fluorescence imaging specifically during gynecologic oncology surgeries involving bowel resections. After surgeons complete the anastomosis, ICG will be administered intravenously. Investigators will then examine the blood flow at the anastomosis site using a special near-infrared camera. If the blood flow appears insufficient, investigators may choose to revise the bowel connection during the same operation.

The study will include approximately 50 women undergoing surgery for gynecologic cancers such as ovarian, uterine, cervical, or vulvar cancer. The primary goal is to determine whether the use of this imaging technique reduces complications, especially within the first 30 days after surgery.

The results of this research could lead to safer surgical procedures, improved patient outcomes, and potentially influence clinical practice guidelines in gynecologic oncology.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older.
* Diagnosis of gynecologic cancer (ovarian, endometrial, cervical, vulvar) requiring surgical treatment.
* Planned bowel resection and anastomosis during gynecologic oncology surgery.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to indocyanine green (ICG).
* Pregnancy or breastfeeding at the time of surgery.
* Severe liver or kidney dysfunction limiting the use of ICG.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are eligible because the study specifically addresses surgical procedures performed for cancers affecting female reproductive organs.
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Anastomotic Complications within 30 Days After Surgery | 30 days after surgery
  The primary outcome will be the incidence of anastomotic leaks, pelvic abscesses, and infections observed within 30 days following bowel anastomosis performed during gynecologic oncology surgery with indocyanine green-enhanced near-infrared fluorescence imaging.

SECONDARY OUTCOMES:
Number of Anastomoses Revised After Indocyanine Green Fluorescence Imaging | Intraoperative (During Surgery)
  The secondary outcome will evaluate how frequently the bowel anastomosis site was revised intraoperatively due to insufficient perfusion as detected by indocyanine green-enhanced near-infrared fluorescence imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Samet Topuz, Prof., Study Chair — Istanbul University; Yagmur Minareci, Assist. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Gynecologic Oncology, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding individual participant data (IPD) sharing has not yet been made. Data sharing will be considered upon completion of the study and publication of results.

REFERENCES:
- [Background] Morales-Conde S, Alarcon I, Yang T, Licardie E, Camacho V, Aguilar Del Castillo F, Balla A. Fluorescence angiography with indocyanine green (ICG) to evaluate anastomosis in colorectal surgery: where does it have more value? Surg Endosc. 2020 Sep;34(9):3897-3907. doi: 10.1007/s00464-019-07159-1. Epub 2019 Oct 4. PMID 31586247
- [Background] Emile SH, Khan SM, Wexner SD. Impact of change in the surgical plan based on indocyanine green fluorescence angiography on the rates of colorectal anastomotic leak: a systematic review and meta-analysis. Surg Endosc. 2022 Apr;36(4):2245-2257. doi: 10.1007/s00464-021-08973-2. Epub 2022 Jan 13. PMID 35024926
- [Background] Chan DKH, Lee SKF, Ang JJ. Indocyanine green fluorescence angiography decreases the risk of colorectal anastomotic leakage: Systematic review and meta-analysis. Surgery. 2020 Dec;168(6):1128-1137. doi: 10.1016/j.surg.2020.08.024. Epub 2020 Oct 1. PMID 33010938
- [Background] Parthasarathy M, Greensmith M, Bowers D, Groot-Wassink T. Risk factors for anastomotic leakage after colorectal resection: a retrospective analysis of 17 518 patients. Colorectal Dis. 2017 Mar;19(3):288-298. doi: 10.1111/codi.13476. PMID 27474844
- [Background] BRUNSCHWIG A. Complete excision of pelvic viscera for advanced carcinoma; a one-stage abdominoperineal operation with end colostomy and bilateral ureteral implantation into the colon above the colostomy. Cancer. 1948 Jul;1(2):177-83. doi: 10.1002/1097-0142(194807)1:23.0.co;2-a. No abstract available. PMID 18875031
- [Background] Grimm C, Harter P, Alesina PF, Prader S, Schneider S, Ataseven B, Meier B, Brunkhorst V, Hinrichs J, Kurzeder C, Heitz F, Kahl A, Traut A, Groeben HT, Walz M, du Bois A. The impact of type and number of bowel resections on anastomotic leakage risk in advanced ovarian cancer surgery. Gynecol Oncol. 2017 Sep;146(3):498-503. doi: 10.1016/j.ygyno.2017.06.007. Epub 2017 Jun 10. PMID 28610745
- [Background] Harter P, Sehouli J, Lorusso D, Reuss A, Vergote I, Marth C, Kim JW, Raspagliesi F, Lampe B, Aletti G, Meier W, Cibula D, Mustea A, Mahner S, Runnebaum IB, Schmalfeldt B, Burges A, Kimmig R, Scambia G, Greggi S, Hilpert F, Hasenburg A, Hillemanns P, Giorda G, von Leffern I, Schade-Brittinger C, Wagner U, du Bois A. A Randomized Trial of Lymphadenectomy in Patients with Advanced Ovarian Neoplasms. N Engl J Med. 2019 Feb 28;380(9):822-832. doi: 10.1056/NEJMoa1808424. PMID 30811909